CLINICAL TRIAL: NCT05331976
Title: A Clinical Evaluation of Proof Diagnostics Test System Including the Proof Diagnostics Reader and COVID-19 Test for Point-of-Care
Brief Title: A Clinical Evaluation of Proof Diagnostics Test System Including the Proof Diagnostics Reader and COVID-19 Test
Status: Completed | Type: Observational
Sponsor: Proof Diagnostics (Industry)
Collaborators: ICON Clinical Research (Industry); MRI Global (Industry); ASCLEPES Research Center (Unknown); Eastside Research Associates (Unknown); PMG Research of Piedmont Healthcare (Unknown)
Responsible Party: Sponsor
Other Study IDs: PDx-2233-01
Record Dates: First submitted 2022-04-14; First posted 2022-04-18 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Asymptomatic COVID-19
Keywords: COVID-19; CRISPR; Diagnostics; Medical Device
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dry anterior nares swabs with self-collected nasal material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic subjects: * Subjects must present with 1 or more signs or symptoms of COVID-19 infection*.
  * Subjects must have experienced symptom onset within the previous 5 days.
  * Subject or Subject's legally authorized representative (LAR) is willing and able to provide informed consent. Adult subjects unable to consent will provide assent in addition to LAR's consent.
  * Subject is ≥ 2 years of age. Subjects 2 ≥ x ≤ 17 will provide assent in addition to parent/legal guardian's consent.
  Interventions: Diagnostic Test: Proof Lab Test System
- Asymptomatic Subjects: * Subject must have been exposed to known SARS-CoV-2 positive or suspected SARS-CoV-2 symptomatic individuals within the previous 5 days.
  * Subject or Subject's legally authorized representative (LAR) is willing and able to provide informed consent. Adult subjects unable to consent will provide assent in addition to LAR's consent.
  * Subject is ≥ 2 years of age. Subjects 2 ≥ x ≤ 17 will provide assent in addition to parent/legal guardian's consent.
  Interventions: Diagnostic Test: Proof Lab Test System

INTERVENTIONS:
Diagnostic Test: Proof Lab Test System — Includes the Proof Lab Reader and the Proof Lab COVID-19 Test Kit containing: Proof Lab COVID-19 Test Cartridge, Sample Vial, Sample Swab, Exact Volume Transfer Pipette

SUMMARY:
To determine the accuracy of Proof Diagnostics COVID-19 Test in the intended, symptomatic and suspected/at-risk asymptomatic population and point-of-care use as compared to a standard molecular comparator, Quidel Lyra SARS-CoV-2 Assay for diagnosing SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The disease was first identified in December 2019 in Wuhan, the capital of China's Hubei province, and has since spread globally, resulting in the ongoing 2019-20 (and now 2021) coronavirus pandemic. The first confirmed case of what was then an unknown coronavirus was traced back to November 2019 in Hubei. Common symptoms include fever, dry cough, fatigue, sputum production, loss of smell, and shortness of breath. While the majority of cases result in mild symptoms, some cases progress to viral pneumonia and multi-organ failure. Emergency symptoms include difficulty breathing, persistent chest pain or pressure, confusion, difficulty waking, and bluish face or lips. The time from exposure to onset of symptoms is typically around five days but may range from two to fourteen days. As of December 4th, 2020, more than 67.3 million cases have been reported across 185 countries and territories, resulting in more than 1.54 million deaths.

On December 2nd, 2020 the Pfizer/BioNTech vaccine was approved in the United Kingdom, followed by approval in the United States (under Emergency Use Authorization [EUA]) on December 11th, 2020. Numerous antiviral and anti-inflammatory treatments have been proposed for COVID-19. Today, management involves the treatment of symptoms, supportive care, isolation, and experimental measures. The WHO has published several testing protocols for the disease. The standard method of testing is real-time reverse transcription polymerase chain reaction (rRT-PCR). The test is typically done on respiratory samples obtained by a nasopharyngeal swab and more recently mid-turbinate and anterior nares nasal swab, and sputum sample or saliva may also be used. Results are generally available within 12-18 hours but can take upwards of two - four days depending on the testing needs of the community. Blood tests can be used, but these require two blood samples taken two weeks apart, and the results have little immediate value. Blood tests can be used to detect antibodies to the virus. The FDA in the United States authorized under EUA the first antigen point-of-care test on 21 March 2020 for use at the end of that month and more recently Lucira has received EUA authorization for at-home-testing.

The FDA has continued to request novel, molecular diagnostic tests which can be offered as point-of-care tests with the potential for future at-home use with a prescription. Proof Diagnostics believes our Proof Diagnostics Test System offers an important improvement to the global testing challenge, providing a state-of-the-art CRISPR-based test for detecting SARS-CoV-2 with sensitivity comparable to the gold standard RT-qPCR (Limit of Detection of ~300 copies/mL, sensitivity >95%, specificity >99%). The Proof Diagnostics Test System thus offers a low-cost and scalable alternative which will be utilized in this clinical study protocol and enable our EUA submission based on the data generated.

ELIGIBILITY:
Inclusion Criteria:

* For Symptomatic Subjects:
* Subjects must present with 1 or more of the following signs or symptoms:

Fever Cough Shortness of Breath Difficulty Breathing Muscle Pain Headache Sore Throat Chills New Loss of Taste or Smell Congestion Runny Nose Diarrhea Nausea or vomiting

* Subjects must have experienced symptom onset within the previous 5 days.
* Subject or Subject's legally authorized representative (LAR) is willing and able to provide informed consent. Adult subjects unable to consent will provide assent in addition to LAR's consent.
* Subject is ≥ 2 years of age. Subjects ages 2 ≥ x ≤ 17 will provide assent in addition to parent/legal guardian's consent.

For Asymptomatic Subjects:

* Asymptomatic subjects must have been exposed to known SARS-CoV-2 positive or suspected SARS-CoV-2 symptomatic individuals within the previous 5 days.
* Subject or Subject's legally authorized representative (LAR) is willing and able to provide informed consent. Adult subjects unable to consent will provide assent in addition to LAR's consent.
* Subject is ≥ 2 years of age. Subjects ages 2 ≥ x ≤ 17 will provide assent in addition to parent/legal guardian's consent.

Note that subjects in recognized vulnerable populations, such as pregnant women and the cognitively impaired, will not be specifically targeted for recruitment, however individual subjects within vulnerable populations may be enrolled. The Human Subject's Protections procedures employed in this protocol are sufficient to protect the rights and welfare of any subject within an eligible vulnerable population and no additional measures are necessary.

Exclusion Criteria:

* The subject is not able to tolerate sample collection.
* The subject has been positive for SARS-CoV-2 previously.
* The subject underwent a nasal wash/aspirate as part of standard of care within 24 hours prior to the study visit.
* The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
* The subject has previously participated in this research study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals exhibiting signs and symptoms of respiratory infection as well as those individuals who are asymptomatic and are suspected of having SARS-CoV-2 or at risk due to exposure to individuals with SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Percent Agreement | Two weeks
  The primary outcome measure will be positive and negative percent agreement (PPA and NPA) of the candidate device in a point-of-care setting to the authorized molecular comparator.

SECONDARY OUTCOMES:
Ratio of Positive Predictive Value to Negative Predictive Value | Two Weeks
  Determine the likelihood ratio of positive predictive value to likelihood ratio negative predictive value, standard positive predictive value, and standard negative predictive value. Additionally, discrepant test results found between the Proof Test and the Quidel Comparator Test will be analyzed via an independent EUA approved test for final adjudication.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Asclepes Research Center, Spring Hill, Florida
  - PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - Eastside Research Associates, Redmond, Washington

IPD SHARING:
Plan to Share IPD: No